CLINICAL TRIAL: NCT06747507
Title: Investigating the Optimal Management of Dolutegravir Resistance: an Open-label Randomised Controlled Trial of Maintaining Dolutegravir or Switch to Ritonavir-boosted Darunavir
Brief Title: Ndovu RCT: Investing the Optimal Management of Dolutegravir Resistance
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Nairobi (Other)
Collaborators: Instituto Nacional de Saúde, Mozambique (Other Government); Muhimbili University of Health and Allied Sciences (Other); SolidarMed (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Loice Achieng Ombajo, Chief Investigator, University of Nairobi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ndovu RCT
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: HIV-1-infection
Keywords: HIV; Dolutegravir; Treatment failure; Drug resistant mutations; Dolutegravir resistance; Re-suppression
MeSH Terms: interventions — dolutegravir

STUDY DESIGN:
Intervention Model Description: This is a phase 3b, multi-country, open-label, two-arm, active-controlled randomized clinical trial over 12 months describing the efficacy and safety of switching from DTG to DRV/r among PLWH age ≥ 3 years who are failing DTG-based ART with HIV-1 RNA ≥ 200 copies/mL and ≥ 1 major DTG-associated DRM (substitution at codon 66K, 92Q, 118R, 138K/A/T, 140S/A/C, 148H/R/K, 155H or 263K ), and most recent prior HIV-1 RNA ≥1,000 copies/mL after at least 6 months on DTG-based ART.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continue on DTG-based Therapy (Experimental): Participants in this arm will continue their pre-randomization DTG-based ART regimen
  Interventions: Drug: Dolutegravir Pill
- Switch to PI-based Therapy (Active Comparator): Participants in this arm will be switched to ritonavir-boosted darunavir (DRV/r)-based ART regimen on the day of randomization
  Interventions: Drug: Darunavir+Ritonavir

INTERVENTIONS:
Drug: Dolutegravir Pill — Dose will be based on weight; brand names will be as supplied through the respective national programs
  Arms: Continue on DTG-based Therapy
Drug: Darunavir+Ritonavir — Dose will be based on weight
  Other Names: Durart
  Arms: Switch to PI-based Therapy

SUMMARY:
This clinical trial will address the gap in published data on the effect of dolutegravir (DTG)-associated drug-resistant mutations on viral suppression among people remaining on DTG-based antiretroviral therapy. It will also address the gap in the optimal management strategy for this population.

DETAILED DESCRIPTION:
BACKGROUND:

The majority of people living with HIV (PLWH) on first-line antiretroviral therapy (ART) in low- and middle-income countries are on dolutegravir (DTG)-containing regimens. Different countries have adopted different approaches in the management of people on DTG-based first-line ART with repeat HIV viral load (VL) of > 1,000 copies/mL after 3 months of enhanced adherence counselling. For example, Kenya recommends a drug resistance test (DRT) to guide on switch and the optimal second-line regimen; Mozambique and Tanzania recommend switch to 2 nucleoside reverse transcriptase inhibitors (NRTIs) and protease inhibitors (PIs) without drug resistance testing; South Africa does not recommend switch from DTG or DRT for those who are on first-line DTG-containing regimens within the first 2 years of treatment, after which management is guided by possible DRT and expert opinion. The World Health Organization has recognised the role of drug resistance testing (DRT) in a treatment failure algorithm for people living with HIV receiving DTG-based treatment to minimise unnecessary switches from this regimen. The switch to PI has disadvantages including higher cost, higher pill burden, less convenient administration (often should be taken with food), more potential drug-drug interactions, poorer tolerability and more long-term toxicities.

GOAL:

To assess the efficacy and safety of remaining on DTG compared to switching to DRV/r among people failing DTG-based ART with at least one major DTG DRM.

METHODS:

This is a phase 3b, multi-country, open-label, two-arm, active-controlled randomized clinical trial (RCT) over 12 months describing the efficacy and safety of switching from DTG to DRV/r among PLWH age ≥ 3 years who are failing DTG-based ART with HIV-1 RNA ≥ 200 copies/mL and ≥ 1 major DTG-associated DRM (and most recent prior HIV-1 RNA ≥ 1,000 copies/mL after at least 6 months on DTG-based ART). The primary efficacy endpoint is the proportion of participants with HIV-1 RNA < 200 copies/mL at month 6. The study will be conducted in 9 sites in Kenya, Mozambique, Tanzania and Lesotho targeting 392 participants including 30 children aged between 3 and 14 years old. The primary efficacy analysis will assess the difference in the proportion of participants with viral suppression at month 6 using the Cochran-Mantel-Haenszel method. This RCT is nested within an observational cohort study describing HIV-1 viral suppression of people with HIV-1 RNA value of ≥ 1,000 copies/mL after at least six months on DTG-based ART.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Ndovu cohort study
* Able and willing to understand and comply with the protocol requirements, instructions and restrictions
* Able and willing to provide informed consent for the nested clinical trial (assent as appropriate and legal guardian consent if < 18 years)
* Age ≥ 3 years
* Most recent HIV-1 RNA ≥ 200 copies/mL
* At least one major DTG-associated DRM (substitution at codon 66K, 92Q, 118R, 138K/A/T, 140S/A/C, 148H/R/K, 155H or 263K)

Exclusion Criteria:

* Pregnant or breastfeeding
* Using any concomitant therapy disallowed as per the reference safety information and product labelling for the study drugs
* WHO stage 3 or 4 opportunistic infection which would prevent randomisation to either arm (e.g. due to drug interactions or significant liver or renal injury) within 4 weeks prior to RCT screening
* Investigator opinion that the potential participant should discontinue DTG immediately for clinical reasons
* Investigator opinion that the potential participant should not switch to DRV/r for clinical reasons

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with HIV-1 RNA of <200 copies/mL at 6 months | 6 months
  The comparative efficacy of switching to a DRV/r-based regimen after confirmed virologic failure and of remaining on DTG-based ART in achieving viral suppression of <200 copies/mL at 6 months from randomization among participants with ≥1 major DTG-associated DRM

SECONDARY OUTCOMES:
Proportion of participants with HIV-1 RNA of <200 copies/mL at 12 months | 12 months
  Viral suppression to HIV-RNA of <200 copies/mL at 12 months from randomization
Superiority of switch to DRV/r | 6 months
  Evaluate if switching to DRV/r-based ART after virologic failure is superior to remaining on DTG-based ART in achieving viral suppression to <200 copies/mL at 6 months from randomization
Viral suppression with cut-off of 50 copies/mL | 6 and 12 months
  Evaluate the difference in viral suppression using HIV-RNA cut-off of <50 copies/mL at 6 and 12 months from randomization
Viral suppression with cut-off of 1,000 copies/mL | 6 and 12 months
  Evaluate the difference in viral suppression using HIV-RNA cut-off of <1,000 copies/mL at 6 and 12 months from randomization
Viral suppression by age strata | 6 and 12 months
  Viral load suppression rate by age strata: 3-9, 10-19, ≥20, 20-24, 25-34, 35-44, and ≥45 years old
Viral suppression by sex at birth | 6 and 12 months
  Viral load suppression based on participant's sex
Incidence of adverse events by study arm | 6 and 12 months
  Incidence and severity of adverse events and laboratory abnormalities
Association between adherence and suppression | 6 months
  Adherence levels, based on DBS TFV-DP levels, associated with suppression and selection of treatment-emergent DRMs
Incidence of drug resistant mutations (DRMs) | 6 and 12 months
  Incidence of treatment-emergent DRMs over 12 months of follow-up
Patterns of accumulated drug resistant mutations (DRMs) | 6 and 12 months
  Describe the patterns of accumulated drug resistant mutations over 12 months of follow-up
Drug resistant mutations (DRM) patterns associated with non-suppression | 6 and 12 months
  Evaluate drug resistant mutation patterns that are associated with sustained non-suppression
Predictors of DTG-associated drug resistant mutations (DRMs) | 6 and 12 months
  Investigate the predictors of selection of DTG-associated drug resistant mutations
Viral suppression by pre-enrolment nucleoside reverse transcriptase inhibitor (NRTI) | 6 and 12 months
  Assess viral suppression based on pre-enrolment NRTI
Viral suppression by tenofovir disoproxil fumarate versus tenofovir alafenamide | 6 and 12 months
  Assess viral suppression based on tenofovir disoproxil fumarate (TDF) versus tenofovir alafenamide (TAF) as the study nucleoside reverse transcriptase inhibitor
Change in cluster of differentiation 4 (CD4) Count | 6 and 12 months
  The impact of regimen on change in cluster of differentiation 4 (CD4) count
Patient satisfaction as measured using the HIV Treatment Satisfaction Questionnaire - Status version (HIVTSQs) which scores 10 variables on a 7-point likert score ranging from 0 to 6 with a higher score representing a better outcome | 6 months
  Patient satisfaction (HIVTSQs) at baseline
Change in patient satisfaction as measured using the HIV Treatment Satisfaction Questionnaire - Change version (HIVTSQc) which scores 10 variables on a 7-point likert score ranging from -3 to +3 with a higher score representing a better outcome | Month 6
  Patient satisfaction (HIVTSQc) at month 6

CONTACTS AND LOCATIONS:
Overall Officials: Loice A Ombajo, MMed, MSc, Principal Investigator — University of Nairobi
Locations (9):
- Kenya (3):
  - Jaramogi Oginga Odinga Teaching and Referral Hospital, Kisumu
  - Bomu Hospital, Mombasa
  - Kenyatta National Hospital, Nairobi
- Lesotho (2):
  - Butha-Buthe District Hospital, Butha-Buthe
  - Mokhotlong District Hospital, Mokhotlong
- Mozambique (3):
  - CS Ponta Gea, Beira, Sofala
  - CS Machava II, Maputo
  - CS Ndlavela, Maputo
- MUHAS Clinical Trial Unit, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share the individual patient data (IPD) that underlie the results reported after de-identification (text, tables, figures and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 6 months after publication of the final manuscript and for a period of 36 months
Access Criteria: Access to IPD will be subject to the University of Nairobi data sharing requirements. Written requests should be submitted to the Chief Investigator providing a brief description of the individual or group making the request and detailing the reason for the same. Prior to sharing the data, the requestor will be required to sign a data access and sharing agreement.